CLINICAL TRIAL: NCT07321262
Title: An Interpretable and Clinically Deployable Machine Learning Model for Predicting Early Postoperative Pneumonia of Brain Tumor: a Multicenter Diagnostic Study
Brief Title: Machine Learning to Predict Postoperative Pneumonia in Brain Tumor Patients
Acronym: ML-PNEUMO-BT
Status: Completed | Type: Observational
Sponsor: Ming Yang (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); Shandong Cancer Hospital and Institute (Other)
Responsible Party: Sponsor-Investigator, Ming Yang, Clinical Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Other Study IDs: NCC2025C-1426; 2024-I2M-3-014 (Other: CAMS Innovation Fund for Medical Sciences)
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pneumonia; Brain Tumors
Keywords: postoperative pneumonia; brain tumor surgery; perioperative management; machine learning; explainable artificial intelligence; SHAP; clinical decision support system
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Retrospective model development cohort (CAMS/PUMC, 2022-2024): Retrospective cohort collected at the Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College (CAMS/PUMC) between Jan 1, 2022 and Oct 31, 2024. Adult patients undergoing elective craniotomy for intracranial brain tumor resection were included. This cohort was used for model development, comparison of candidate algorithms, and internal validation; it was randomly split 8:2 into a training set (n=609) and an internal validation set (n=152). Early postoperative pneumonia (POP) was defined by CDC criteria within 7 days postoperatively. No study-mandated intervention was applied; routine perioperative care was provided.
- Prospective internal validation cohort (Test P, CAMS/PUMC): Prospective cohort enrolled at CAMS/PUMC between Nov 1, 2024 and Apr 30, 2025 (Test P; n=224). Adult patients undergoing elective craniotomy for brain tumor resection were included. This cohort prospectively validated the finalized interpretable prediction model for early POP using routinely available perioperative EMR variables. Early POP was defined per CDC criteria within 7 postoperative days. Clinical management followed standard-of-care without any study-assigned intervention.
- Prospective external validation cohort (Test A, Anhui Medical Univ): Prospective external validation cohort recruited at the First Affiliated Hospital of Anhui Medical University from Aug 1, 2024 to Apr 30, 2025 (Test A; n=329). Adult patients undergoing elective craniotomy for brain tumor resection were included. The cohort independently validated the finalized POP prediction model using routine perioperative data. Early POP was defined by CDC criteria within 7 days after surgery. No investigational intervention was administered; all care followed local standard practice.
- Prospective external validation cohort (Test S, Shandong Cancer Hospital): Prospective external validation cohort recruited at Shandong Cancer Hospital from Aug 1, 2024 to Apr 30, 2025 (Test S; n=440). Adult patients undergoing elective craniotomy for intracranial brain tumor resection were included. This cohort was used to externally validate the finalized interpretable model for early POP prediction using routinely collected perioperative variables. Early POP was defined according to CDC criteria within 7 postoperative days. Participants received routine perioperative management per institutional standards without study-mandated interventions.
- Prospective external validation cohort (Test J, Jinan Fourth People's Hospital): Prospective external validation cohort recruited at Jinan Fourth People's Hospital from Aug 1, 2024 to Apr 30, 2025 (Test J; n=102). Adult patients undergoing elective craniotomy for brain tumor resection were included. The cohort externally validated the finalized prediction model for early POP based on routine perioperative EMR data. Early POP was defined per CDC criteria within 7 postoperative days. There was no study-assigned intervention; all patients received standard perioperative care per local protocols.

SUMMARY:
Postoperative pneumonia (POP) is a common and serious complication after elective craniotomy for brain tumor resection. POP often develops within the first week after surgery and may lead to prolonged hospitalization, higher medical costs, and increased risk of severe illness. Because symptoms can be subtle in neurosurgical patients, POP may be detected late, limiting timely prevention and treatment.

This study will evaluate whether a machine-learning-based clinical decision support tool can help clinicians identify patients at high risk for POP early and improve perioperative preventive care. The tool uses routinely collected clinical information to estimate an individual patient's POP risk and provides an easy-to-understand explanation of key risk drivers. Based on the predicted risk level (low, moderate, high, or very high), the system suggests standardized preventive care pathways (e.g., perioperative airway management, targeted antibiotic strategies per local practice, and nutritional support), while allowing clinicians to override recommendations at any time.

Participants will be adults undergoing their first elective craniotomy for brain tumor resection at participating neurosurgical centers. The primary outcome is the occurrence of POP within 7 days after surgery, defined using CDC/NHSN criteria. Secondary outcomes include antibiotic use intensity, length of hospital stay, direct medical cost, and clinician decision confidence. Participants will be followed at postoperative days 1, 3, and 7 using electronic medical record review and phone confirmation when needed.

The goal of this study is to determine whether integrating an explainable AI risk prediction tool into routine care can reduce POP and improve the quality and efficiency of perioperative management after brain tumor surgery.

DETAILED DESCRIPTION:
Rationale Postoperative pneumonia (POP) remains a frequent and clinically important complication after elective craniotomy for brain tumor resection, contributing to prolonged hospitalization, increased cost, and worse clinical outcomes. Conventional POP risk assessment is often experience-based or relies on simplified scoring approaches, which may not adequately capture nonlinear interactions among perioperative factors. This study implements an explainable machine-learning (ML) prediction model within routine perioperative workflows and evaluates whether model-assisted care can improve POP prevention and related resource utilization compared with usual care.

Decision support system

An explainable gradient boosting machine (GBM) model is used to estimate individual POP risk from routinely available perioperative variables. Interpretability is provided using SHAP-based explanations at two complementary levels:

Population level: summarizes the most influential predictors and selected interaction patterns to support clinical understanding and model governance.

Patient level: generates an individualized contribution visualization (e.g., waterfall-style), highlighting the main drivers of a specific patient's risk estimate.

The system automatically assigns a risk tier (low, moderate, high, or very high) and links each tier to standardized prevention pathway templates (e.g., airway management optimization, antimicrobial stewardship-consistent strategies per local policy, and nutritional support). The tool does not mandate treatment; clinicians may accept, modify, or override any suggestion.

Evaluation framework The overall project includes retrospective model development/optimization, prospective external validation/calibration, and a pragmatic implementation evaluation. The registered interventional evaluation uses a multicenter, cluster randomized crossover design with monthly alternating periods of model-assisted care versus usual care. Allocation procedures, eligibility criteria, planned enrollment, and endpoint definitions/time windows are specified in the corresponding record modules (Study Design, Arms/Interventions, Outcome Measures, and Eligibility) to avoid duplication in this section.

Implementation and integration The model is deployed as a lightweight web service with unified APIs and data-exchange formats to enable non-disruptive integration with hospital information systems (HIS) and electronic medical records (EMR). A web-based front end and a Python-based back end support RESTful calls and are designed for low-latency inference (target single-prediction latency <200 ms), suitable for perioperative and inpatient workflows.

Data governance and model updating To support long-term generalizability across hospitals and mitigate dataset shift, the project establishes a closed-loop maintenance process ("local de-identification → cloud retraining → model version management → edge deployment"). Model updates are version-controlled and deployed under governance procedures consistent with local regulations, institutional policies, and applicable ethics approvals.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Undergoing elective craniotomy for intracranial brain tumor resection.
* Perioperative clinical data available in the electronic medical record to derive required predictors.
* Expected postoperative survival ≥ 7 days.

Exclusion Criteria:

* Evidence of active infection (including pneumonia) prior to surgery.
* Thoracic surgery or severe chest trauma within 30 days prior to craniotomy.
* Spinal tumors or extracranial peripheral nerve tumors.
* Pregnancy or lactation.
* Hospice care, expected survival < 7 days, or insufficient data completeness for model calculation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective craniotomy for intracranial brain tumor resection at participating centers. The study includes a retrospective model-development cohort and multiple prospective validation cohorts. Routinely collected perioperative electronic medical record data are used to develop and validate an interpretable prediction model for early postoperative pneumonia (within 7 postoperative days).
Sampling Method: Non-Probability Sample
Enrollment: 1856 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of early postoperative pneumonia (POP) | Within 7 days after craniotomy (postoperative day 0-7)
  Early POP was diagnosed according to CDC criteria and recorded in the electronic medical record, assessed as a binary outcome (POP vs no POP) within 7 postoperative days.

SECONDARY OUTCOMES:
Discrimination of the finalized prediction model (AUC) | Within 7 days after craniotomy (postoperative day 0-7)
  Area under the receiver operating characteristic curve (AUC) for the finalized interpretable logistic regression model in predicting early POP (binary outcome within 7 days).
Calibration performance of the finalized prediction model | Within 7 days after craniotomy (postoperative day 0-7)
  Calibration assessed using calibration curve and summary statistics (e.g., calibration intercept and slope; Brier score), comparing predicted probabilities with observed early POP outcomes.
Clinical utility of the finalized prediction model (Decision Curve Analysis) | Within 7 days after craniotomy (postoperative day 0-7)
  Net benefit of the finalized model evaluated by decision curve analysis across clinically relevant threshold probabilities for early POP.
Classification performance of the finalized prediction model at a pre-specified cutoff | Within 7 days after craniotomy (postoperative day 0-7)
  Sensitivity, specificity, accuracy, positive predictive value (PPV), negative predictive value (NPV), and F1 score calculated at a pre-specified probability threshold (e.g., determined in the training cohort using Youden index) and applied to validation cohorts.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing is currently undecided. The study uses detailed multi-center electronic medical record data, and additional assessment is needed to determine whether an adequately de-identified dataset can be shared without meaningful risk of re-identification and in compliance with IRB/ethics approvals, institutional policies, and applicable privacy regulations. We will revisit the IPD sharing plan after study completion and publication of primary results.

REFERENCES:
- [Background] Lundberg SM, Lee S-I. A unified approach to interpreting model predictions. Advances in Neural Information Processing Systems. 2017;30
- [Background] Azodi CB, Tang J, Shiu SH. Opening the Black Box: Interpretable Machine Learning for Geneticists. Trends Genet. 2020 Jun;36(6):442-455. doi: 10.1016/j.tig.2020.03.005. Epub 2020 Apr 17. PMID 32396837
- [Background] Han J, Yao T, Gao L, Gao H, Chen Y, Wang Y, Cao Y, Liu C, Qiu F, Jia K, Huang H. Development and validation of a risk prediction model related to inflammatory and nutritional indexes for postoperative pulmonary infection after radical colorectal cancer surgery. BMJ Open. 2025 Jan 8;15(1):e087426. doi: 10.1136/bmjopen-2024-087426. PMID 39779267
- [Background] Zhao C, Xiang B, Zhang J, Yang P, Liu Q, Wang S. Predicting postoperative pulmonary infection risk in patients with diabetes using machine learning. Front Physiol. 2024 Dec 4;15:1501854. doi: 10.3389/fphys.2024.1501854. eCollection 2024. PMID 39697615
- [Background] Chen Y, Ma M, Qu D, Xu C. Machine learning and transformer models for prediction of postoperative pneumonia risk in patients with lower limb fractures. Sci Rep. 2025 Jul 1;15(1):22409. doi: 10.1038/s41598-025-04623-y. PMID 40595785
- [Background] Churpek MM, Carey KA, Edelson DP, Singh T, Astor BC, Gilbert ER, Winslow C, Shah N, Afshar M, Koyner JL. Internal and External Validation of a Machine Learning Risk Score for Acute Kidney Injury. JAMA Netw Open. 2020 Aug 3;3(8):e2012892. doi: 10.1001/jamanetworkopen.2020.12892. PMID 32780123
- [Background] Koyner JL, Adhikari R, Edelson DP, Churpek MM. Development of a Multicenter Ward-Based AKI Prediction Model. Clin J Am Soc Nephrol. 2016 Nov 7;11(11):1935-1943. doi: 10.2215/CJN.00280116. Epub 2016 Sep 15. PMID 27633727
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Lan J, Wei Y, Zhu Y, Zhang Y, Zhang S, Mo L, Wei D, Lei Y. Risk Factors for Post-Operative Pulmonary Infection in Patients With Brain Tumors: A Systematic Review and Meta-Analysis. Surg Infect (Larchmt). 2023 Sep;24(7):588-597. doi: 10.1089/sur.2023.130. Epub 2023 Aug 10. PMID 37582199
- [Background] Jing X, Wang X, Zhuang H, Fang X, Xu H. Multiple Machine Learning Approaches Based on Postoperative Prediction of Pulmonary Complications in Patients With Emergency Cerebral Hemorrhage Surgery. Front Surg. 2022 Jan 18;8:797872. doi: 10.3389/fsurg.2021.797872. eCollection 2021. PMID 35127804
- [Background] Sughrue ME, Rutkowski MJ, Shangari G, Chang HQ, Parsa AT, Berger MS, McDermott MW. Risk factors for the development of serious medical complications after resection of meningiomas. Clinical article. J Neurosurg. 2011 Mar;114(3):697-704. doi: 10.3171/2010.6.JNS091974. Epub 2010 Jul 23. PMID 20653395
- [Background] Longo M, Agarwal V. Postoperative Pulmonary Complications Following Brain Tumor Resection: A National Database Analysis. World Neurosurg. 2019 Jun;126:e1147-e1154. doi: 10.1016/j.wneu.2019.03.058. Epub 2019 Mar 15. PMID 30880210
- [Background] Gonzalez-Bonet LG, Tarazona-Santabalbina FJ, Lizan Tudela L. [Neurosurgery in the elderly patient: Geriatric neurosurgery]. Neurocirugia (Astur). 2016 Jul-Aug;27(4):155-66. doi: 10.1016/j.neucir.2015.11.003. Epub 2016 Jan 4. Spanish. PMID 26762658
- [Background] Karhade AV, Cote DJ, Larsen AM, Smith TR. Neurosurgical Infection Rates and Risk Factors: A National Surgical Quality Improvement Program Analysis of 132,000 Patients, 2006-2014. World Neurosurg. 2017 Jan;97:205-212. doi: 10.1016/j.wneu.2016.09.056. Epub 2016 Sep 23. PMID 27671880
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] Lan J, Liu X, Mo L, Wei D, Zhang S, Zhang Y, Zhu Y, Lei Y. Construction and validation of a risk prediction model for postoperative pulmonary infection in patients with brain tumor: a retrospective study. PeerJ. 2025 Mar 31;13:e18996. doi: 10.7717/peerj.18996. eCollection 2025. PMID 40183067